CLINICAL TRIAL: NCT01267422
Title: Safety and Efficacy Study of a Single Intravitreal Injection of rAAV2-ND4 Treatment of Leber Hereditary Optic Neuropathy
Brief Title: Safety and Efficacy Study of rAAV2-ND4 Treatment of Leber Hereditary Optic Neuropathy (LHON)
Acronym: rAAV2-ND4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bin Li (Other)
Collaborators: Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor-Investigator, Bin Li, Safety and Efficacy Study of rAAV2-ND4 Treatment of LHON, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAVCT-2
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Leber Hereditary Optic Neuropathy
Keywords: Leber's Hereditary Optic Neuropathy,11778 LHON mutation,; rAAV2-ND4,triamcinolone acetonide
MeSH Terms: conditions — Optic Atrophy, Hereditary, Leber

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rAAV2-ND4 (Experimental): injection
  Interventions: Drug: rAAV2-ND4

INTERVENTIONS:
Drug: rAAV2-ND4 — injection
  Other Names: rAAV2-ND4 gene therapy

SUMMARY:
This study is meant to assess the safety and efficacy of rAAV2-ND4 treatment of Leber hereditary optic neuropathy with 11778 LHON mutation.

DETAILED DESCRIPTION:
Leber's Hereditary Optic Neuropathy (LHON) is a maternally inherited ocular disorder associated with a mutation in mtDNA . The common manifestation is visual loss which caused by the respiratory chain enzymes complex dysfunction resulting in increased oxidative stress enzymes production.

Material and Method Seven patients with 11778 LHON mutation were randomly treated with a Single IVT Injection of recombinant Adeno-Associated Virus-NADH dehydrogenase, subunit 4 (complex I)（rAAV2-ND4)（0.05ml).The dose was 5 × 10^9 vg/0.05 mL for patients younger than 12 years old, and 1 × 10^10 vg/0.05 mL for patients older than 12 years old. The visual acuity, visual evoked potential （VEP）,optical coherence tomography（ OCT）, computerized visual field, electroretinograms(ERG), retinal nerve fiber layer(RNFL)and Liver and kidney function in plasma were compared before and after treatment at 1,3,and 6, months interval.

ELIGIBILITY:
Inclusion Criteria:

1. comply with Leber hereditary optic neuropathy diagnostic criteria.
2. in patients with informed consent, voluntary participation.
3. signed informed consent.
4. 8 ≤ Age ≤ 60 years old, good health, the patient can tolerate local anesthesia surgery.
5. to comply with doctor's instructions, can in the time of referral.

Exclusion Criteria:

1. Cardiopulmonary and renal function in severe weakness, cancer, a variety of bleeding disorders, acute sensing disease, high fever, high fever disease, women during pregnancy, heart disease, such as post-operative recovery period.
2. Are participating in other clinical studies of patients.
3. Patients with mental disorders.

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2011-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: bin Li, PhD,MD, Study Chair — Deputy Director of Ophthalmology
Locations (1):
- Department of Ophthalmology ，Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carelli V, Ross-Cisneros FN, Sadun AA. Mitochondrial dysfunction as a cause of optic neuropathies. Prog Retin Eye Res. 2004 Jan;23(1):53-89. doi: 10.1016/j.preteyeres.2003.10.003. PMID 14766317
- [Background] Mackey DA, Oostra RJ, Rosenberg T, Nikoskelainen E, Bronte-Stewart J, Poulton J, Harding AE, Govan G, Bolhuis PA, Norby S. Primary pathogenic mtDNA mutations in multigeneration pedigrees with Leber hereditary optic neuropathy. Am J Hum Genet. 1996 Aug;59(2):481-5. No abstract available. PMID 8755941
- [Background] Wallace DC, Singh G, Lott MT, Hodge JA, Schurr TG, Lezza AM, Elsas LJ 2nd, Nikoskelainen EK. Mitochondrial DNA mutation associated with Leber's hereditary optic neuropathy. Science. 1988 Dec 9;242(4884):1427-30. doi: 10.1126/science.3201231.
- [Background] Oguchi Y. [Past, present, and future in Leber's hereditary optic neuropathy]. Nippon Ganka Gakkai Zasshi. 2001 Dec;105(12):809-27. Japanese. PMID 11802455
- [Background] Cui G, Ding H, Xu Y, Li B, Wang DW. Applications of the method of high resolution melting analysis for diagnosis of Leber's disease and the three primary mutation spectrum of LHON in the Han Chinese population. Gene. 2013 Jan 1;512(1):108-12. doi: 10.1016/j.gene.2012.09.110. Epub 2012 Oct 9. PMID 23063736
- [Background] Mashima Y, Kigasawa K, Wakakura M, Oguchi Y. Do idebenone and vitamin therapy shorten the time to achieve visual recovery in Leber hereditary optic neuropathy? J Neuroophthalmol. 2000 Sep;20(3):166-70. doi: 10.1097/00041327-200020030-00006. PMID 11001192
- [Background] Carelli V, Barboni P, Zacchini A, Mancini R, Monari L, Cevoli S, Liguori R, Sensi M, Lugaresi E, Montagna P. Leber's Hereditary Optic Neuropathy (LHON) with 14484/ND6 mutation in a North African patient. J Neurol Sci. 1998 Oct 8;160(2):183-8. doi: 10.1016/s0022-510x(98)00239-1. PMID 9849804
- [Background] Barnils N, Mesa E, Munoz S, Ferrer-Artola A, Arruga J. [Response to idebenone and multivitamin therapy in Leber's hereditary optic neuropathy]. Arch Soc Esp Oftalmol. 2007 Jun;82(6):377-80. doi: 10.4321/s0365-66912007000600012. Spanish. PMID 17573650
- [Background] Angebault C, Gueguen N, Desquiret-Dumas V, Chevrollier A, Guillet V, Verny C, Cassereau J, Ferre M, Milea D, Amati-Bonneau P, Bonneau D, Procaccio V, Reynier P, Loiseau D. Idebenone increases mitochondrial complex I activity in fibroblasts from LHON patients while producing contradictory effects on respiration. BMC Res Notes. 2011 Dec 22;4:557. doi: 10.1186/1756-0500-4-557. PMID 22192149
- [Background] Klopstock T, Yu-Wai-Man P, Dimitriadis K, Rouleau J, Heck S, Bailie M, Atawan A, Chattopadhyay S, Schubert M, Garip A, Kernt M, Petraki D, Rummey C, Leinonen M, Metz G, Griffiths PG, Meier T, Chinnery PF. A randomized placebo-controlled trial of idebenone in Leber's hereditary optic neuropathy. Brain. 2011 Sep;134(Pt 9):2677-86. doi: 10.1093/brain/awr170. Epub 2011 Jul 25. PMID 21788663
- [Background] Carelli V, La Morgia C, Valentino ML, Rizzo G, Carbonelli M, De Negri AM, Sadun F, Carta A, Guerriero S, Simonelli F, Sadun AA, Aggarwal D, Liguori R, Avoni P, Baruzzi A, Zeviani M, Montagna P, Barboni P. Idebenone treatment in Leber's hereditary optic neuropathy. Brain. 2011 Sep;134(Pt 9):e188. doi: 10.1093/brain/awr180. Epub 2011 Aug 2. No abstract available. PMID 21810891
- [Background] Sadun AA, Chicani CF, Ross-Cisneros FN, Barboni P, Thoolen M, Shrader WD, Kubis K, Carelli V, Miller G. Effect of EPI-743 on the clinical course of the mitochondrial disease Leber hereditary optic neuropathy. Arch Neurol. 2012 Mar;69(3):331-8. doi: 10.1001/archneurol.2011.2972. PMID 22410442
- [Background] Newman NJ. Treatment of Leber hereditary optic neuropathy. Brain. 2011 Sep;134(Pt 9):2447-50. doi: 10.1093/brain/awr192. Epub 2011 Aug 22. No abstract available. PMID 21859767
- [Background] Maguire AM, Simonelli F, Pierce EA, Pugh EN Jr, Mingozzi F, Bennicelli J, Banfi S, Marshall KA, Testa F, Surace EM, Rossi S, Lyubarsky A, Arruda VR, Konkle B, Stone E, Sun J, Jacobs J, Dell'Osso L, Hertle R, Ma JX, Redmond TM, Zhu X, Hauck B, Zelenaia O, Shindler KS, Maguire MG, Wright JF, Volpe NJ, McDonnell JW, Auricchio A, High KA, Bennett J. Safety and efficacy of gene transfer for Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2240-8. doi: 10.1056/NEJMoa0802315. Epub 2008 Apr 27. PMID 18441370
- [Background] Bainbridge JW, Smith AJ, Barker SS, Robbie S, Henderson R, Balaggan K, Viswanathan A, Holder GE, Stockman A, Tyler N, Petersen-Jones S, Bhattacharya SS, Thrasher AJ, Fitzke FW, Carter BJ, Rubin GS, Moore AT, Ali RR. Effect of gene therapy on visual function in Leber's congenital amaurosis. N Engl J Med. 2008 May 22;358(21):2231-9. doi: 10.1056/NEJMoa0802268. Epub 2008 Apr 27. PMID 18441371
- [Background] Bonnet C, Kaltimbacher V, Ellouze S, Augustin S, Benit P, Forster V, Rustin P, Sahel JA, Corral-Debrinski M. Allotopic mRNA localization to the mitochondrial surface rescues respiratory chain defects in fibroblasts harboring mitochondrial DNA mutations affecting complex I or v subunits. Rejuvenation Res. 2007 Jun;10(2):127-44. doi: 10.1089/rej.2006.0526. PMID 17518546
- [Background] Ellouze S, Augustin S, Bouaita A, Bonnet C, Simonutti M, Forster V, Picaud S, Sahel JA, Corral-Debrinski M. Optimized allotopic expression of the human mitochondrial ND4 prevents blindness in a rat model of mitochondrial dysfunction. Am J Hum Genet. 2008 Sep;83(3):373-87. doi: 10.1016/j.ajhg.2008.08.013. Epub 2008 Sep 4. PMID 18771762
- [Background] Koilkonda RD, Yu H, Chou TH, Feuer WJ, Ruggeri M, Porciatti V, Tse D, Hauswirth WW, Chiodo V, Boye SL, Lewin AS, Neuringer M, Renner L, Guy J. Safety and effects of the vector for the Leber hereditary optic neuropathy gene therapy clinical trial. JAMA Ophthalmol. 2014 Apr 1;132(4):409-20. doi: 10.1001/jamaophthalmol.2013.7630. PMID 24457989
- [Background] Koilkonda R, Yu H, Talla V, Porciatti V, Feuer WJ, Hauswirth WW, Chiodo V, Erger KE, Boye SL, Lewin AS, Conlon TJ, Renner L, Neuringer M, Detrisac C, Guy J. LHON gene therapy vector prevents visual loss and optic neuropathy induced by G11778A mutant mitochondrial DNA: biodistribution and toxicology profile. Invest Ophthalmol Vis Sci. 2014 Oct 23;55(12):7739-53. doi: 10.1167/iovs.14-15388. PMID 25342621
- [Background] Shi H, Gao J, Pei H, Liu R, Hu WK, Wan X, Li T, Li B. Adeno-associated virus-mediated gene delivery of the human ND4 complex I subunit in rabbit eyes. Clin Exp Ophthalmol. 2012 Dec;40(9):888-94. doi: 10.1111/j.1442-9071.2012.02815.x. Epub 2012 Jul 2. PMID 22612072
- [Background] Mays LE, Vandenberghe LH, Xiao R, Bell P, Nam HJ, Agbandje-McKenna M, Wilson JM. Adeno-associated virus capsid structure drives CD4-dependent CD8+ T cell response to vector encoded proteins. J Immunol. 2009 May 15;182(10):6051-60. doi: 10.4049/jimmunol.0803965. PMID 19414756
- [Background] Hsu TK, Wang AG, Yen MY, Liu JH. Leber's hereditary optic neuropathy masquerading as optic neuritis with spontaneous visual recovery. Clin Exp Optom. 2014 Jan;97(1):84-6. doi: 10.1111/cxo.12100. Epub 2013 Aug 1. PMID 23905692
- [Background] Leo-Kottler B, Christ-Adler M. [Leber optic neuropathy in women and children]. Ophthalmologe. 1999 Nov;96(11):698-701. doi: 10.1007/s003470050479. German. PMID 10631830
- [Background] Li H, Tuyishime S, Wu TL, Giles-Davis W, Zhou D, Xiao W, High KA, Ertl HC. Adeno-associated virus vectors serotype 2 induce prolonged proliferation of capsid-specific CD8+ T cells in mice. Mol Ther. 2011 Mar;19(3):536-46. doi: 10.1038/mt.2010.267. Epub 2010 Dec 14. PMID 21157435
- [Background] Giordano C, Montopoli M, Perli E, Orlandi M, Fantin M, Ross-Cisneros FN, Caparrotta L, Martinuzzi A, Ragazzi E, Ghelli A, Sadun AA, d'Amati G, Carelli V. Oestrogens ameliorate mitochondrial dysfunction in Leber's hereditary optic neuropathy. Brain. 2011 Jan;134(Pt 1):220-34. doi: 10.1093/brain/awq276. Epub 2010 Oct 13. PMID 20943885
- [Background] Testa F, Maguire AM, Rossi S, Pierce EA, Melillo P, Marshall K, Banfi S, Surace EM, Sun J, Acerra C, Wright JF, Wellman J, High KA, Auricchio A, Bennett J, Simonelli F. Three-year follow-up after unilateral subretinal delivery of adeno-associated virus in patients with Leber congenital Amaurosis type 2. Ophthalmology. 2013 Jun;120(6):1283-91. doi: 10.1016/j.ophtha.2012.11.048. Epub 2013 Mar 6. PMID 23474247
- [Background] Yang S, He H, Zhu Y, Wan X, Zhou LF, Wang J, Wang WF, Liu L, Li B. Chemical and material communication between the optic nerves in rats. Clin Exp Ophthalmol. 2015 Nov;43(8):742-8. doi: 10.1111/ceo.12547. Epub 2015 Jun 25. PMID 25950380
- [Background] Ghelli A, Porcelli AM, Zanna C, Martinuzzi A, Carelli V, Rugolo M. Protection against oxidant-induced apoptosis by exogenous glutathione in Leber hereditary optic neuropathy cybrids. Invest Ophthalmol Vis Sci. 2008 Feb;49(2):671-6. doi: 10.1167/iovs.07-0880. PMID 18235013
- [Background] Yu-Wai-Man P, Griffiths PG, Chinnery PF. Mitochondrial optic neuropathies - disease mechanisms and therapeutic strategies. Prog Retin Eye Res. 2011 Mar;30(2):81-114. doi: 10.1016/j.preteyeres.2010.11.002. Epub 2010 Nov 26. PMID 21112411
- [Background] Koilkonda RD, Guy J. Leber's Hereditary Optic Neuropathy-Gene Therapy: From Benchtop to Bedside. J Ophthalmol. 2011;2011:179412. doi: 10.1155/2011/179412. Epub 2010 Dec 26. PMID 21253496
- [Result] Wan X, Pei H, Zhao MJ, Yang S, Hu WK, He H, Ma SQ, Zhang G, Dong XY, Chen C, Wang DW, Li B. Efficacy and Safety of rAAV2-ND4 Treatment for Leber's Hereditary Optic Neuropathy. Sci Rep. 2016 Feb 19;6:21587. doi: 10.1038/srep21587. PMID 26892229
- [Derived] Liu HL, Yuan JJ, Tian Z, Li X, Song L, Li B. What are the characteristics and progression of visual field defects in patients with Leber hereditary optic neuropathy: a prospective single-centre study in China. BMJ Open. 2019 Mar 15;9(3):e025307. doi: 10.1136/bmjopen-2018-025307. PMID 30878986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients diagnosed with LHON (with a verified point mutation at the 11778 nucleotide site)
Pre-assignment Details: All patients were administered rAAV2-ND4 by intravitreal injection to one eye and then followed for 36 months.
Groups:
- Participants Receiving Treatment in Left Eye: 5 participants receiving treatment in left eye
- Participants Receiving Treatment in Right Eye: 4 participants receiving treatment in right eye
Period: Intravitreal rAAV2-ND4 Injection
Arm/Group | Participants Receiving Treatment in Left Eye | Participants Receiving Treatment in Right Eye
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0
Period: Safety and Efficacy Study
Arm/Group | Participants Receiving Treatment in Left Eye | Participants Receiving Treatment in Right Eye
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Age,Gender,Ethnicity,Race,Region of Enrollment
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15 [7.65 to 30.79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 9

OUTCOME MEASURES:

1. Primary Outcome: The Best Corrected Visual Acuity(BCVA)
Time Frame: Up to 3 years
Population: The data are expressed as mean±standard error. Comparisons before and after treatment of the BCVA were analyzed using the paired t-test.A probability (P) value of less than 0.05 was considered statistically significant.Lower logMAR represents a better outcome.
Measure: Mean (Standard Error); unit: logMAR
Units Other Than Participants: logMAR
Groups:
- BCVA of Un-treated Eyes: BCVA of un-treated eyes in 9 patients
- BCVA of Treated Eyes: BCVA of trearted eyes in 9 patients
Arm/Group | BCVA of Un-treated Eyes | BCVA of Treated Eyes
Number analyzed (Participants) | 9 | 9
Number analyzed (logMAR) | 9 | 9
logMAR
  before treament | 1.40 (0.55) | 1.69 (0.43)
  1 months after treament | 1.36 (0.58) | 1.58 (0.44)
  3 months after treament | 1.31 (0.58) | 1.38 (0.46)
  6 months after treament | 1.20 (0.68) | 1.23 (0.60)
  9 months after treament | 1.23 (0.62) | 1.27 (0.58)

2. Primary Outcome: Results of CD3/CD4/CD8 Test
Description: The mean percentage of CD3+/CD4+/CD8+ test before and after treatment
Time Frame: up to 6 months
Measure: Mean (Full Range); unit: Percentage of total cells
Groups:
- The Mean Percentage of CD3+/CD4+/CD8+ Before Treatment: The mean percentage of CD3+ before treatment;The mean percentage of CD4+ before treatment;The mean percentage of CD8+ before treatment
- The Mean Percentage of CD3+/CD4+/CD8+ After Treatment: The mean percentage of CD3+ after treatment;The mean percentage of CD4+ after treatment;The mean percentage of CD8+ after treatment
Arm/Group | The Mean Percentage of CD3+/CD4+/CD8+ Before Treatment | The Mean Percentage of CD3+/CD4+/CD8+ After Treatment
Number analyzed (Participants) | 9 | 9
Percentage of total cells
  Values of CD3+ | 51 [50 to 84] | 53 [50 to 84]
  Values of CD4+ | 26 [20 to 51] | 20 [20 to 51]
  Values of CD8+ | 20 [12 to 45] | 13 [12 to 45]

3. Secondary Outcome: Intraocular Pressure;
Time Frame: Up to 3 years
Measure: Mean (Full Range); unit: mmHg
Groups:
- IOP Before Treatment: Ophthalmologic examinations includes IOP of 9 paticipants before treatment
- IOP After Treatment: Ophthalmologic examinations includes IOP of 9 participants after treatment
Arm/Group | IOP Before Treatment | IOP After Treatment
Number analyzed (Participants) | 9 | 9
mmHg | 14 [10 to 21] | 16 [10 to 21]

4. Secondary Outcome: Neutralizing Antibody Assay
Description: The mean of Neutralizing antibody assay of 8 patients before and after treatment
Time Frame: up to 3 years
Population: Neutralizing antibody assay of 8 patients except Patient 1 because he once accepted the other eye's treatment
Measure: Mean (Standard Deviation); unit: titer
Groups:
- The Mean of Neutralizing Antibody Assay Before Treatment: The mean of Neutralizing antibody assay before treatment of 8 patients
- The Mean of Neutralizing Antibody Assay After Treatment: The mean of Neutralizing antibody assay after treatment of 8 patients
Arm/Group | The Mean of Neutralizing Antibody Assay Before Treatment | The Mean of Neutralizing Antibody Assay After Treatment
Number analyzed (Participants) | 8 | 8
titer | 0.9221 (0.142437) | 0.8723 (0.201054)

5. Secondary Outcome: Average RNFL Thickness Througth Optical Coherence Tomography(OCT) Test
Description: Average RNFL thickness of 8 patients througth Optical coherence tomography(OCT) test before and after treatment
Time Frame: Up to 3 years
Population: RNFL thickness of 8 patients except Patient 1 because he once accepted the other eye's treatment
Measure: Mean (Standard Deviation); unit: Micrometer
Groups:
- Average RNFL Thickness Before Treatment: Average RNFL thickness before treatment of injected eyes;Average RNFL thickness before treatment of uninjected eyes
- Average RNFL Thickness After Treatment: Average RNFL thickness after treatment of injected eyes;Average RNFL thickness after treatment of uninjected eyes
Arm/Group | Average RNFL Thickness Before Treatment | Average RNFL Thickness After Treatment
Number analyzed (Participants) | 8 | 8
Micrometer
  injected eye | 47.3125 (7.87259) | 46.7813 (7.5397)
  uninjected eye | 50.1875 (13.402) | 47.9688 (9.7031)

6. Secondary Outcome: Computerized Visual Field(MD: Mean Deviation, the Value Close to 0 Regarded Normal)
Description: MD: mean deviation, the value Close to 0 regarded normal.VFI/MD：The bigger one was more close to the normal value.
Time Frame: up to 3 years
Population: Patient 2 refused the vision field test,there are MD outcome measure of 8 patients.
Measure: Mean (Standard Deviation); unit: dB
Groups:
- Mean MD Before Treatment: Mean MD before treatment of injected eyes;Mean MD before treatment of uninjected eyes
- Mean MD After Treatment: Mean MD after treatment of injected eyes;Mean MD after treatment of uninjected eyes
Arm/Group | Mean MD Before Treatment | Mean MD After Treatment
Number analyzed (Participants) | 8 | 8
dB
  injected eye | -29.377 (5.16805) | -23.813 (7.27537)
  uninjected eye | -28.701 (3.65595) | -23.427 (8.15747)

7. Secondary Outcome: Computerized Visual Field(VFI: Visual Field Index ,the Value Close to 100% Regarded Normal)
Description: VFI: visual field index ,the value Close to 100% regarded normal. VFI/MD：The bigger one was more close to the normal value.
Time Frame: up to 3 years
Population: Patient 2 refused the vision field test,there are VFI outcome measure of 8 patients.
Measure: Mean (Standard Deviation); unit: Percentage of normal
Groups:
- Mean VFI Before Treatment: Mean VFI before treatment of injected eyes;Mean VFI before treatment of uninjected eyes
- Mean VFI After Treatment: Mean VFI after treatment of injected eyes;Mean VFI after treatment of uninjected eyes
Arm/Group | Mean VFI Before Treatment | Mean VFI After Treatment
Number analyzed (Participants) | 8 | 8
Percentage of normal
  injected eye | 11 (0.14513) | 28 (0.23305)
  uninjected eye | 10.5 (0.28714) | 25 (0.24804)

ADVERSE EVENTS:
Groups:
- Short-term Affects: Lens may be injured during intravitreal injection, and cataract is probably complicated. Retinal detachment or endophthalmitis may be complicated due to retina injury.IOP raised.Endophthalmitis after treament. Hyper-susceptibility or immune response during surgery or after surgery.
- Long-term Affects: Lens may be injured after intravitreal injection, and cataract is probably complicated. Retinal detachment or endophthalmitis may be complicated due to retina injury.IOP raised.Blood and urine routine is affected.Liver and kidney function is affected.Immune response after surgery.
Arm/Group | Short-term Affects | Long-term Affects
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No